CLINICAL TRIAL: NCT01392560
Title: An Open-label 8-week Adjunctive-to-insulin and Renal Mechanistic Pilot Trial of BI 10773 in Type 1 Diabetes Mellitus (the ATIRMA Trial)
Brief Title: Safety and Efficacy of Empagliflozin (BI 10773) in Type 1 Diabetes Mellitus Patients With or Without Renal Hyperfiltration
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1245.46
Record Dates: First submitted 2011-07-11; First posted 2011-07-12 (Estimated); Results first posted 2014-06-17 (Estimated); Last update posted 2014-06-17 (Estimated); Status verified 2014-05

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — empagliflozin

ARMS (1):
- BI 10773 (Experimental): Oral once daily
  Interventions: Drug: BI 10773

INTERVENTIONS:
Drug: BI 10773 — Oral once daily

SUMMARY:
This open-label study aims to evaluate the impact of BI 10773 treatment on glomerular filtration rate under controlled conditions of euglycaemia and hyperglycaemia in subjects with type 1 diabetes mellitus with or without renal hyperfiltration and to characterize the safety and efficacy of BI 10773 25 mg QD as add-on therapy to insulin in these subjects.

ELIGIBILITY:
Inclusion criteria:

1. Male or female subjects 18 years of age or older diagnosed with type 1 diabetes mellitus
2. Glycated hemoglobin (HbA1C) of 6.5% to 11.0% and an estimated glomerular filtration rate (eGFR) greater or equal to 60 ml/min/1.73m² at screening
3. Subjects must be either experienced insulin pump users or be on multiple daily injections of any type of insulin

Exclusion criteria:

1. Evidence of macroalbuminuria or leukocyte positive urinalysis at screening
2. Any concomitant medication known to interfere with renin-angiotensin-aldosterone system (RAAS) activity or treatment with any other drugs to reduce blood glucose other than insulin
3. History of macrovascular disease or any other disease which would interfere with trial participation or any ongoing clinical condition that would jeopardize subject safety or study compliance based on investigator judgement

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2011-06; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- 1245.46.10001 Boehringer Ingelheim Investigational Site, Toronto, Ontario, Canada

REFERENCES:
- [Derived] van Bommel EJM, Lytvyn Y, Perkins BA, Soleymanlou N, Fagan NM, Koitka-Weber A, Joles JA, Cherney DZI, van Raalte DH. Renal hemodynamic effects of sodium-glucose cotransporter 2 inhibitors in hyperfiltering people with type 1 diabetes and people with type 2 diabetes and normal kidney function. Kidney Int. 2020 Apr;97(4):631-635. doi: 10.1016/j.kint.2019.12.021. No abstract available. PMID 32200854
- [Derived] Perkins BA, Cherney DZ, Soleymanlou N, Lee JA, Partridge H, Tschirhart H, Zinman B, Mazze R, Fagan N, Kaspers S, Woerle HJ, Broedl UC, Johansen OE. Diurnal Glycemic Patterns during an 8-Week Open-Label Proof-of-Concept Trial of Empagliflozin in Type 1 Diabetes. PLoS One. 2015 Nov 6;10(11):e0141085. doi: 10.1371/journal.pone.0141085. eCollection 2015. PMID 26544192
- [Derived] Perkins BA, Cherney DZ, Partridge H, Soleymanlou N, Tschirhart H, Zinman B, Fagan NM, Kaspers S, Woerle HJ, Broedl UC, Johansen OE. Sodium-glucose cotransporter 2 inhibition and glycemic control in type 1 diabetes: results of an 8-week open-label proof-of-concept trial. Diabetes Care. 2014 May;37(5):1480-3. doi: 10.2337/dc13-2338. Epub 2014 Mar 4. PMID 24595630
- [Derived] Cherney DZ, Perkins BA, Soleymanlou N, Har R, Fagan N, Johansen OE, Woerle HJ, von Eynatten M, Broedl UC. The effect of empagliflozin on arterial stiffness and heart rate variability in subjects with uncomplicated type 1 diabetes mellitus. Cardiovasc Diabetol. 2014 Jan 29;13:28. doi: 10.1186/1475-2840-13-28. PMID 24475922
- [Derived] Cherney DZ, Perkins BA, Soleymanlou N, Maione M, Lai V, Lee A, Fagan NM, Woerle HJ, Johansen OE, Broedl UC, von Eynatten M. Renal hemodynamic effect of sodium-glucose cotransporter 2 inhibition in patients with type 1 diabetes mellitus. Circulation. 2014 Feb 4;129(5):587-97. doi: 10.1161/CIRCULATIONAHA.113.005081. Epub 2013 Dec 13. PMID 24334175

RESULTS

PARTICIPANT FLOW:
Groups:
- Empagliflozin (BI 10773) 25 mg: Oral once daily
  Empagliflozin 25 mg: Oral once daily
Period: Overall Study
Arm/Group | Empagliflozin (BI 10773) 25 mg
Started | 52
Completed | 40
Not Completed | 12
Not completed — Adverse Event | 2
Not completed — not entered | 8
Not completed — discontinued during placebo run-in | 2

BASELINE CHARACTERISTICS:
Population: Treated Set
Arm/Group | Empagliflozin (BI 10773) 25 mg
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.1 (5.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22
  Male | 20

OUTCOME MEASURES:

1. Primary Outcome: Change in Glomerular Filtration Rate (GFR) After 8 Weeks of Treatment With Empagliflozin Under Controlled Conditions of Euglycaemia and Hyperglycaemia
Description: The primary endpoint is change in glomerular filtration rate (GFR) after 8 weeks of treatment with empagliflozin under controlled conditions of euglycaemia and hyperglycaemia
Time Frame: Baseline and 8 weeks
Population: Per protocol set for renal (PPS_RENAL) consists of all patients who were treated with study drug and had a baseline measurement and evaluable post-dosing renal data under the clamped hyperglycemia condition for the primary endpoint.
Measure: Mean (Standard Error); unit: mL/min/1.73 m^2
Groups:
- All Patients (Empagliflozin 25 mg): All patients (hyperfilterers and non-hyperfilterers)
  Empagliflozin 25 mg: Oral once daily
- Hyperfilterers (Empagliflozin 25 mg): Hyperfilterers
  Empagliflozin 25 mg: Oral once daily
  hyperfilterers = GFRs of ≥135 mL/min/1.73m2
- Non-hyperfilterers (Empagliflozin 25 mg): Non-hyperfilterers
  Empagliflozin 25 mg: Oral once daily
  non-hyperfilterers = GFRs of ≥60 mL/min/1.73m2 to <135 mL/min/1.73m2
Arm/Group | All Patients (Empagliflozin 25 mg) | Hyperfilterers (Empagliflozin 25 mg) | Non-hyperfilterers (Empagliflozin 25 mg)
Number analyzed (Participants) | 40 | 27 | 13
mL/min/1.73 m^2
  Euglycaemia | -19.6 (5.6) | -33.4 (6.2) | 9.0 (5.9)
  Hyperglycaemia | -30.8 (6.2) | -44.5 (7.1) | -2.4 (7.7)
Statistical Analysis 1: Comparison: All Patients (Empagliflozin 25 mg); Test of the difference between baseline and end of treatment under euglycaemia condition for all patients; Test type: Superiority or Other; p = 0.0011, Paired t-test; Mean change from baseline = -19.6, Standard Error of Mean 5.6 — Estimated value = mean of end of treatment - baseline
Statistical Analysis 2: Comparison: All Patients (Empagliflozin 25 mg); Test the difference between baseline and end of treatment under hyperglycaemia condition for all patients; Test type: Superiority or Other; p < 0.0001, Paired t-test; Mean change from baseline = -30.8, Standard Error of Mean 6.2 — Estimated value = mean of end of treatment - baseline
Statistical Analysis 3: Comparison: Hyperfilterers (Empagliflozin 25 mg); Test of the difference between baseline and end of treatment under euglycaemia condition for hyperfilterers; Test type: Superiority or Other; p < 0.0001, Paired t-test; Change from baseline = -33.4, Standard Error of Mean 6.2 — Estimated value = mean of end of treatment - baseline
Statistical Analysis 4: Comparison: Hyperfilterers (Empagliflozin 25 mg); Test of the difference between baseline and end of treatment under hyperglycaemia condition for hyperfilterers; Test type: Superiority or Other; p < 0.0001, Paired t-test; Mean change from baseline = -44.5, Standard Error of Mean 7.1 — Estimated value = mean of end of treatment - baseline
Statistical Analysis 5: Comparison: Non-hyperfilterers (Empagliflozin 25 mg); Test of the difference between baseline and end of treatment under euglycaemia condition for non-hyperfilterers; Test type: Superiority or Other; p = 0.1524, Paired t-test; Mean change from baseline = 9.0, Standard Error of Mean 5.9 — Estimated value = mean of end of treatment - baseline
Statistical Analysis 6: Comparison: Non-hyperfilterers (Empagliflozin 25 mg); Test of the difference between baseline and end of treatment under hyperglycaemia condition for non-filterers; Test type: Superiority or Other; p = 0.7585, Paired t-test; Mean change from baseline = -2.4, Standard Error of Mean 7.7 — Estimated value = mean of end of treatment - baseline

ADVERSE EVENTS:
Time Frame: 8 weeks
Description: All adverse events, serious and non-serious, occurring during the course of the clinical trial were to be collected, documented and reported to the sponsor by the investigator on the appropriate case reporting forms. Reporting was performed according to the specific definitions and instructions.
Groups:
- Empagliflozin 25 mg: Oral once daily
  Empagliflozin 25 mg: Oral once daily
Arm/Group | Empagliflozin 25 mg
Serious Adverse Events (participants affected / at risk) | 3/42
Other Adverse Events (participants affected / at risk) | 42/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 25 mg (N=42)
Gastroenteritis viral (Infections and infestations) | 1
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Empagliflozin 25 mg (N=42)
Abdominal pain (Gastrointestinal disorders) | 5
Dry mouth (Gastrointestinal disorders) | 7
Nausea (Gastrointestinal disorders) | 7
Vomiting (Gastrointestinal disorders) | 6
Thirst (General disorders) | 31
Genitourinary tract infection (Infections and infestations) | 6
Influenza (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 40
Back pain (Musculoskeletal and connective tissue disorders) | 4
Dizziness (Nervous system disorders) | 6
Headache (Nervous system disorders) | 10
Pollakiuria (Renal and urinary disorders) | 33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.